CLINICAL TRIAL: NCT01137929
Title: Bacterial and Host Genetic Risk Factors That Predispose Children to Acute Pyelonephritis and Renal Scarring
Brief Title: Bacterial and Host Genetic Risk Factors in Acute Pyelonephritis
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty identifying eligible candidates
Sponsor: Hans Pohl (Other)
Responsible Party: Sponsor-Investigator, Hans Pohl, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: Genes-APN
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Vesicoureteral Reflux
Keywords: Vesicoureteral reflux; Kidney; Renal Scar; Urinary tract infection
MeSH Terms: conditions — Vesico-Ureteral Reflux; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples: Urine is routinely collected at the time of presentation with fever to diagnose UTI and an aliquot of this urine sample will be frozen for microbial genomic and metagenomic sequencing and analysis, that will allow us to identify unique/pathogenic/virulence factors in the genomes of these bacterial species when compared to non-pathogenic strains that have been subject to whole genome sequencing.
  Blood: DNA samples will be obtained at the time of renal scanning from the study subjects. The genomic DNA is used in PCR reactions and the resulting PCR products are screened for single nucelotide polymorphisms. Although we will be performing a genome wide association study, we will be particularly curious as to the behavior of SNP's among certain previously described candidates for the risk of renal scarring such as TLR2, TLR4, TGF-beta, and TNF-alpha. DNA samples will be stored for possible use in other future association studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- With APN, With VUR, With Renal Scar: This group of children who present with a febrile UTI will be found to have APN on DMSA renal scan and will also have VUR by VCUG and a renal scar on follow-up DMSA renal scan.
- With APN, With VUR, Without Renal Scar: This group of children who present with a febrile UTI will be found to have APN on DMSA renal scan and will also have VUR by VCUG and NO renal scar on follow-up DMSA renal scan.
- With APN, without VUR, with Renal Scar: This group of children who present with a febrile UTI will be found to have APN on DMSA renal scan but who will NOT have VUR by VCUG; however they will have a renal scar on follow-up DMSA renal scan.
- With APN, Without VUR, Without Renal Scar: This group of children who present with a febrile UTI will be found to have APN on DMSA renal scan and will NOT have VUR by VCUG, NOR will they have a renal scar on follow-up DMSA renal scan.
- Without APN, With VUR: This group of children who present with a febrile UTI will be found NOT to have APN on DMSA renal scan and will also have VUR by VCUG. They will not undergo a second DMSA scan since the first one is normal.
- Without APN, Without VUR: This group of children who present with a febrile UTI will be found NOT to have APN on DMSA renal scan and will also NOT have VUR by VCUG, NOR a renal scar on follow-up DMSA renal scan.

SUMMARY:
No single host or pathogen trait identified by previous research can be correlated with all cases of childhood acute pyelonephritis or APN (i.e., kidney/upper urinary tract infections) and APN-associated renal scarring (the outcome with the highest morbidity), making it difficult for physicians to determine which patients will be affected. Our proposal is to comprehensively study the relationships between the clinical manifestations of urinary tract infections (UTIs), the host risk factors and immune response, and the microbial species that cause these conditions. The result of the study will be a clinical severity score to personalize diagnostic and treatment strategies for infants with UTI, with the goal of decreasing the morbidity of APN/renal scarring and improving patient outcomes.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are the most common serious bacterial infections in young children, with acute pyelonephritis or APN (i.e., kidney/upper urinary tract infections) and APN-associated renal scarring causing the most potential long-term damage to a child's health. Approximately two-thirds of young children with febrile UTI (UTIF or UTI presenting with fever) will have APN, making UTIF a major indicator of APN. Other than the presence of fever, it is currently difficult for physicians to determine which infant patients have or will develop APN and renal scarring. Individual risk factors for the host (e.g., uncircumcised males, cytokine production) and the pathogen (e.g., presence of fimbriae for adhesion) have individually been linked to APN and renal scarring, but no single trait identified can be correlated with all cases. Multiple factors on both sides of the host-pathogen relationship likely interact to determine the severity of the illness and the outcome. Although the NIDDK/NIH is currently funding two clinical trials to investigate the rate of recurrent UTI and the rate of renal scarring in children (Randomized Intervention of Children with Vesicoureteral REflux, RIVUR; and Careful urinary Tract Infection Evaluation, CUTIE) neither of these studies will be able to identify the child's initial risk for having APN since patient recruitment will occur too long after treatment of the UTI. Also, neither study proposes as a specific goal to obtain bacteriological samples with which to study the microbe's role in the pathogenesis of APN. Thus, to the best of our knowledge, no comprehensive study exists that aims to analyze the relationships between the clinical manifestations of UTIs, the host risk factors and immune response, and the microbial species that cause these conditions. Our proposed collaborative study between Children's National Medical Center (CNMC) and the J. Craig Venter Institute (JCVI) will collect clinical data as well as urine and blood samples from six distinct infant patient populations presenting with UTIF and correlate the clinical, host, and pathogen data for each patient with the severity of the disease and development of APN and renal scarring. Metagenomic and genomic sequencing on the urine and isolated bacteria, respectively, will allow us to comprehensively study both the culturable and unculturable pathogens responsible for the UTI. Using a genome-wide association study (GWAS) we will evaluate the polymorphisms of all known UTI-associated host genes, paying particular attention to the immune system host genes previously identified as potentially linked to APN. To correlate all collected data a publicly available database and website will be created to allow physicians and scientists to traverse the data. Using the data collected in the database, the final result of the study will be a clinical severity score to personalize diagnostic and treatment strategies for infants with UTIF, with the goal of decreasing the morbidity of APN and improving patient outcomes. An improved understanding of the microbial risk factors associated with APN and renal scarring will allow for better diagnostic approaches and improved methods for treating patients, inclusive of novel medications in at risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the inpatient ward at Children's National Medical Center for the treatment of a febrile urinary tract infection (see definitions) will be screened for inclusion into the research protocol.
* UTIF: A UTIF will require the presence of

  * (1) fever and/or symptoms consistent with UTI,
  * (2) pyuria based on urinalysis, and
  * (3) culture-proven infection with a single organism. Specifically, the study definition of UTIF will require:
* Fever: A documented temperature of at least 100.4 °F or 38°C, measured anywhere on the body either at home or at doctor's office.

Positive dipstick analysis: Pyuria on urinalysis (>10 WBC/mm3 (uncentrifuged specimen) OR >5 WBC/hpf (centrifuged specimen), OR >1+ leukocyte esterase on dipstick).

* Culture documentation of UTI: Evidence of bacteria (>5 x 104 CFU/mL (catheterized or suprapubic aspiration urine specimen). Bag collected specimens will not be acceptable

Exclusion Criteria:

* Infants who do not conform to the above inclusion criteria and who have co-morbidities such as duplication abnormalities, diabetes mellitus, over weight status, anatomical defects of the urinary tract and neuropathic bladder dysfunction.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will identify infants ≤ 2 years to be of particular risk for UTIF and renal scarring by virtue of a variety of risk factors, including age, gender, race, and underlying genetic risk factors and bacterial phenotypes.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute pyelonephritis lesions | < 72 hours after presentation with fever and positive urine culture
  Children under two years of age will undergo a 99m-Tc-DMSA renal scan for the detection of acute pyelonephritis lesions within 72 hours of presentation to the ED for evaluation of a fever and positive urine culture. Based on finding the characteristic lesions (such as preservation of the renal contour but with diminished photopenia.
  This outcome measure will be aggregated with other bacterial and host related risk factors in order to identify the salient ones that result in morbidity from bladder infection.

SECONDARY OUTCOMES:
Incidence of renal cortical scarring | At least 6 months
  Since the lesions associated with acute pyelonephritis can resolve up to 6 months following infection, we will stress the importance of obtaining these delayed scans for the purpose of ascertaining whether the inflammation has resulted in a fixed lesion, termed a renal scar.